CLINICAL TRIAL: NCT04835753
Title: Effects Of Extracorporeal Shock Wave On Spastic Equines Foot In Children With Hemiplegic Cerebral Palsy
Brief Title: Shock Wave and Spastic Cerebral Palsy Equines Foot
Acronym: CP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taibah University (Other)
Responsible Party: Principal Investigator, Hatem Abd Elmohsen Abdel Hamid Emara, DR, Taibah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: taibah university
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Extracorporeal Shock Wave Therapy; Hemiplegia; selective motor control
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): received the traditional physical therapy program as muscle stretching and strengthening and neurodevelopmental techniques, proprioceptive training, and balance and gait training plus shock wave on the muscle belly of the planter flexor hypertonic muscles.
  Interventions: Device: shock wave; Other: traditional physical therapy program
- control group (Other): received the traditional physical therapy program as muscle stretching and strengthening and neurodevelopmental techniques, proprioceptive training, and balance and gait training .these traditional therapy had been approved by previous studies its effectiveness in management cerebral palsy child
  Interventions: Other: traditional physical therapy program

INTERVENTIONS:
Device: shock wave — true radial ESWT.A rESW pneumatic device (SHOCK MED, Italy) was used to provide one session per week (for a total of 12-week)
  Arms: study group
Other: traditional physical therapy program — lower limbs muscles stretch and strength in addition to balance and gait training

SUMMARY:
A double-blind randomized controlled study was carried out on 34 children (19 boys and 15 girls) in the age ranged from 7 to 9 years old with spastic hemiplegia were randomly allocated to one of two groups: control or study group. The two groups received traditional therapeutic exercises for 12 weeks. Additionally, study group received rESW (one session/week) on gastrocnemius and soleus muscles (1500 shots/muscle, frequency of 4Hz, energy of 0.030 mJ/mm2). All children were evaluated at baseline, and after 12 weeks by Modified Ashworth Scale, Biodex system 4 isokinetic dynamometer, Gross Motor Function Measure (GMFM-88), dimensions "D" standing and "E" walking, Trost Selective Motor Control Test, and Single Leg Standing Test.

DETAILED DESCRIPTION:
Both groups underwent conventional physical therapy program which included muscle stretching, strengthening exercises, neurodevelopmental techniques, proprioceptive training, and balance and gait training for three months (3 days/week ,1 hour/day).

Study group Subjects in this group received the traditional physical therapy treatment plus true radial ESWT.A rESW pneumatic device (SHOCK MED, Italy) was used to provide one session per week (for a total of 12-week) of shock wave intervention. The pressure pulses were focused on the muscle belly of the planter flexor hypertonic muscles. Standard ultrasonic gel was used as a contact medium. A total of 1500 shots with a pressure of 1.5 bar and an energy flux density (EFD) of 0.030 mJ/mm2 were applied with the repetition frequency of shock wave irradiation of 4 pulses per second (Hz). The rESW session lasted about 6 minutes and was painless; thus, local anesthesia was not required.

ELIGIBILITY:
Inclusion Criteria:

* 1) children who could walk independently or with assistive devices ,2) children with motor dysfunction graded as a 1 or 2 on the Gross Motor Function Classification System (GMFCS), 3) children scoring 1or1+ on the Modified Ashworth Scale (MAS), 4) Dynamic ankle contracture which was confirmed if ankle equinus was observed during ambulation and passive dorsiflexion of the ankle could be accomplished beyond the neutral position with knee extended

Exclusion Criteria:

* 1) children older than 9 years or younger than 7 years, 2) previous botulinum toxin type A injection in the gastrocnemius muscle or serial casting of the ankle within 6 months prior to enrollment, 3) fixed ankle contracture, and 4) surgery of the lower limbs in the past 12 months.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
Biodex system | 12 weeks
  The Biodex system 4 (Biodex Medical, Shirley, NY, USA) was used for the quantitative biomechanical assessment of the spasticity of the affected side ankle plantar flexor muscle
The modified Ashworth scale | 12 weeks
  The modified Ashworth scale, which is a six-point ordinal scale for grading (0, 1, 1+, 2, 3, and 4) was applied for clinical assessment of spasticity of ankle plantar flexors.
Single Leg Standing Test (SLS) | 12 weeks
  The SLS is a simple and effective test to assess static balance. It is conducted by measuring the time that a child can maintain balance by lifting the foot according to the signal "Start." The average of three measures was used.
The Trost Selective Motor Control test (TSMC) | 12 weeks
  The TSMC test was used to assess ability of the child to perform isolated movement of the ankle.

CONTACTS AND LOCATIONS:
Overall Officials: hatem emaraa, PHD, Principal Investigator — Taibah University,saudi arabia
Locations (1):
- Taibah University, Al Madīnah, Saudi Arabia